CLINICAL TRIAL: NCT01792284
Title: A Comparison of LY2605541 Once Daily at a Fixed Time With LY2605541 Variable Time of Dosing in Participants With Type 1 Diabetes Mellitus: An Open Label, Randomized, Crossover Study
Brief Title: A Study of LY2605541 in Participants With Type 1 Diabetes Mellitus
Acronym: IMAGINE 7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14184; I2R-MC-BIAX (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — LY2605541; basal insulin peglispro; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2605541 Fixed Time Dosing (Experimental): Participant-specific dose of LY2605541 administered subcutaneously (SQ) at approximately the same time every evening for 12 weeks in the Lead-in Period and in Randomization Period 1 or Randomization Period 2.
  Participant-specific dose of insulin lispro SQ when >20% of calories were consumed (pre-meal).
  Insulin dose and adjustments to insulin dose were determined by insulin algorithms based on self-monitored blood glucose (SMBG). Target glucose values were as follows:
  Preprandial and bedtime BG between 71 and 130 milligrams/deciliter (mg/dL) Insulin adjustment and glucose correction between 71 and 100 mg/dL.
  Interventions: Drug: LY2605541; Drug: Insulin Lispro
- LY2605541 Variable Time Dosing (Experimental): Participant-specific dose of LY2605541 administered SQ on a variable time schedule (8- and 40-hour dosing intervals) for 12 weeks in Randomization Period 1 or Randomization Period 2. Dosing schedules were to remain approximately the same throughout the 12 weeks.
  Participant-specific dose of insulin lispro SQ when >20% of calories were consumed (pre-meal).
  Insulin dose and adjustments to insulin dose were determined by insulin algorithms based on SMBG. Target glucose values were as follows:
  Preprandial and bedtime BG between 71 and 130 mg/dL Insulin adjustment and glucose correction between 71 and 100 mg/dL.
  Interventions: Drug: LY2605541; Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY2605541
  Other Names: Insulin Peglispro
Drug: Insulin Lispro — All participants will be administering insulin lispro SQ as their pre-meal insulin during the course of the trial.

SUMMARY:
The primary purpose of participation in this study is to compare the safety and efficacy of different dosing schedules of LY2605541 and how different dosing schedules of LY2605541 affect Hemoglobin A1c (HbA1c). Participants will be treated for up to 36 weeks with LY2605541 (one 12-week Lead-in period and two 12-week Randomization periods) and will participate in a total of 42 weeks of total study enrollment, including a 2-week Screening period and a 4-week Follow-up period.

DETAILED DESCRIPTION:
This study involved a comparison of LY2605541 regimens, each administered with bolus insulin lispro. Eligible participants were switched to a fixed evening LY2605541dosing regimen at the beginning of the 12-week lead-in period. LY2605541 was administered SQ once-daily using a prefilled insulin device. The LY2605541dose was adjusted using a dosing algorithm adapted from Bartley and Bolli (Bartley et al. 2008, Bolli et al. 2009) based on the participant's blood glucose (BG) values and documented hypoglycemia during the previous week. Participants not already receiving insulin lispro for prandial dosing were switched to insulin lispro at the beginning of the 12-week lead-in period. Adjustments to insulin lispro doses were based on the insulin dosing algorithms adapted from Riddle and Bergenstal (Riddle et al. 2003, Bergenstal et al. 2008). At the time of randomization, participants were randomized to begin either the fixed evening dosing regimen or the variable time dosing regimen. Each participant was crossed over to the alternate regimen after 12 weeks. The insulin device (prefilled pen) remained the same throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for at least 1 year
* Have an HbA1c value <9.0%
* Have a body mass index (BMI) ≤35.0 kilogram per square meter (kg/m^2)
* Currently using basal/ bolus insulin
* Women of childbearing potential are not breastfeeding and must use methods to prevent pregnancy

Exclusion Criteria:

* Have excessive insulin resistance
* Are taking medications other than insulin for diabetes
* High triglycerides
* Have had more than 1 episode of severe hypoglycemia (defined as requiring assistance due to neurologically disabling hypoglycemia as determined by the investigator) within 6 months prior to entry into the study
* Have had 2 or more emergency room visits or hospitalizations due to poor glucose control (hyperglycemia or diabetic ketoacidosis) in the past 6 months
* Have cardiac disease with functional status that is New York Heart Association (NYHA) Class III or IV (per NYHA Cardiac Disease Classification)
* Have impaired renal function
* Have impaired liver function
* Have had a blood transfusion or severe blood loss within 3 months prior to screening or have known hemoglobinopathy, hemolytic anemia, sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with HbA1c measurement
* Have cancer, recent cancer, or risk of cancer
* Have a known hypersensitivity or allergy to any of the study insulins or their excipients
* Have chronic systemic glucocorticoid users
* Have clinically significant diabetic autonomic neuropathy
* Have irregular sleep/wake cycle
* Have been treated with a drug within the last 30 days that has not received regulatory approval at the time of study entry
* Prior study participation
* Are using or have used niacin preparations as a lipid-lowering medication and/or bile acid sequestrants within 90 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (18):
- United States (17):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aurora, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roswell, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Crystal Lake, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Round Rock, Texas
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayamón, Puerto Rico

REFERENCES:
- [Derived] Qu Y, White RD, Ruberg SJ. Accurate Collection of Reasons for Treatment Discontinuation to Better Define Estimands in Clinical Trials. Ther Innov Regul Sci. 2023 May;57(3):521-528. doi: 10.1007/s43441-022-00491-0. Epub 2022 Dec 21. PMID 36542287

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed a 12 week (wk) Lead-in Period during which insulin peglispro was administered at fixed time in the evening. Participants were then randomized to a fixed evening dose regimen or a variable time dose regimen for 12 wks (Randomization Period 1); after 12 wks, they crossed over to the alternate regimen (Randomization Period 2).
Groups:
- LY2605541 Fixed Time Dosing (All Participants): Lead-in Period: Participant-specific dose of LY2605541 administered subcutaneously (SQ) at approximately the same time every evening for 12 weeks. Participant-specific dose of insulin lispro SQ when >20% of calories were consumed (pre-meal).
  Insulin dose and adjustments to insulin dose were determined by insulin algorithms based on self-monitored blood glucose (SMBG).
  Target glucose values were as follows:
  Preprandial and bedtime BG between 71 and 130 milligrams/deciliter (mg/dL) Insulin adjustment and glucose correction between 71 and 100 mg/dL.
- LY2605541 Fixed Time Dosing, LY2605541 Variable Time Dosing: Randomization Period 1: Participant-specific dose of LY2605541 administered SQ at approximately the same time every evening for 12 weeks. Participant-specific dose of insulin lispro SQ when >20% of calories were consumed (pre-meal).
  Randomization Period 2: Participant-specific dose of LY2605541 administered SQ on a variable schedule (8- and 40-hour dosing intervals) for 12 weeks. Participants were dosed in the morning on Monday, Wednesday, and Friday and in the evening on Tuesday, Thursday, Saturday, and Sunday. Dosing schedules were to remain approximately the same throughout the 12 weeks. Participant-specific dose of insulin lispro SQ when >20% of calories were consumed (pre-meal).
  Insulin dose and adjustments to insulin dose were determined by insulin algorithms based on SMBG. Target glucose values were as follows:
  Preprandial and bedtime BG between 71 and 130 mg/dL Insulin adjustment and glucose correction between 71 and 100 mg/dL.
- LY2605541 Variable Time Dosing, LY2605541 Fixed Time Dosing: Randomization Period 1: Participant-specific dose of LY2605541 administered SQ on a variable schedule (8- and 40-hour dosing intervals) for 12 weeks. Participants were dosed in the morning on Monday, Wednesday, and Friday and in the evening on Tuesday, Thursday, Saturday, and Sunday. Dosing schedules were to remain approximately the same throughout the 12 weeks. Participant-specific dose of insulin lispro SQ when >20% of calories were consumed (pre-meal).
  Randomization Period 2: Participant-specific dose of LY2605541 administered SQ at approximately the same time every evening for 12 weeks. Participant-specific dose of insulin lispro SQ when >20% of calories were consumed (pre-meal).
  Insulin dose and adjustments to insulin dose were determined by insulin algorithms based on SMBG. Target glucose values were as follows:
  Preprandial and bedtime BG between 71 and 130 mg/dL Insulin adjustment and glucose correction between 71 and 100 mg/dL.
Period: Lead-in Period
Arm/Group | LY2605541 Fixed Time Dosing (All Participants) | LY2605541 Fixed Time Dosing, LY2605541 Variable Time Dosing | LY2605541 Variable Time Dosing, LY2605541 Fixed Time Dosing
Started | 212 | 0 | 0
Completed | 182 (Participants that completed the Lead-in Period were randomized and entered Randomization Period 1.) | 0 | 0
Not Completed | 30 | 0 | 0
Not completed — Adverse Event | 15 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Required Discontinuation | 1 | 0 | 0
Period: Randomization Period 1
Arm/Group | LY2605541 Fixed Time Dosing (All Participants) | LY2605541 Fixed Time Dosing, LY2605541 Variable Time Dosing | LY2605541 Variable Time Dosing, LY2605541 Fixed Time Dosing
Started | 0 | 92 | 90
Received at Least 1 Dose of Study Drug | 0 | 92 | 90
Completed | 0 | 90 | 85
Not Completed | 0 | 2 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Period: Randomization Period 2
Arm/Group | LY2605541 Fixed Time Dosing (All Participants) | LY2605541 Fixed Time Dosing, LY2605541 Variable Time Dosing | LY2605541 Variable Time Dosing, LY2605541 Fixed Time Dosing
Started | 0 | 90 | 85
Received at Least 1 Dose of Study Drug | 0 | 90 | 85
Completed | 0 | 87 | 85
Not Completed | 0 | 3 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- All Enrolled Participants: Participants entered a 12-week Lead-in Period where they received fixed time of dose of LY2605541 with bolus insulin lispro. Participants were then randomized to either a fixed time of dose or a variable time of dose regimen for 12 weeks administered with bolus insulin lispro; after 12 weeks, they crossed over to the alternate regimen. LY2605541 dose was adjusted using a dosing algorithm based on the participant's BG values and documented hypoglycemia during the previous week. Insulin dose were determined by insulin algorithms based on SMBG.
  Fixed time of dose: Participant-specific dose of LY2605541 administered SQ at approximately the same time every evening for 12 weeks administered with bolus insulin lispro.
  Variable time of dose: Participant-specific dose of LY2605541 administered SQ on a variable schedule (8- and 40-hour dosing intervals) for 12 weeks. Dosing schedules were to remain approximately the same throughout the 12 weeks administered with bolus insulin lispro.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.08 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98
  Male | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26
  Not Hispanic or Latino | 186
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 203
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 199
  Puerto Rico | 13

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c) at 12 Weeks
Description: HbA1c is a test that measures a person's average blood glucose level over the past 2 to 3 months. Least Squares (LS) means were calculated using a mixed model repeated measures (MMRM) analysis including the following fixed effects: treatment, period, sequence, baseline HbA1c (last nonmissing value at or before randomization), week (defined from the start of each Randomization Period), and treatment-by-week interaction.
Time Frame: At 12 Week in Each Randomization Period
Population: Participants who were randomized, received at least 1 dose of study drug after randomization, and had evaluable HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- LY2605541 Fixed Time Dosing: Participant-specific dose of LY2605541 administered SQ at approximately the same time every evening for 12 weeks.
- LY2605541 Variable Time Dosing: Participant-specific dose of LY2605541 administered SQ on a variable schedule (8- and 40-hour dosing intervals) for 12 weeks. Dosing schedules were to remain approximately the same throughout the 12 weeks.
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 171 | 180
percentage of HbA1c | 6.87 (0.04) | 6.93 (0.04)

2. Secondary Outcome: 30-Day Adjusted Rate of Total and Nocturnal Hypoglycemic Events
Description: Total hypoglycemic events (HE) include any event based on a blood glucose <=70 milligrams per deciliter (mg/dL) (3.9 millimoles per liter [mmol/L]), with or without signs/symptoms of hypoglycemia or an event associated with signs/symptoms of hypoglycemia but without a glucose measurement. Nocturnal HE include any total HE that occurred between bedtime and waking. Group Means are presented and were calculated from negative binomial regression models (number of episodes = treatment + period + treatment sequence + baseline HbA1c [<=8.0% or >8.0%], with log [exposure in days/30] as an offset variable). Group Mean (LS mean) is estimated by taking the inverse link function on individual participant covariates first and then averages over all participants.
Time Frame: Baseline (Day 1) of Randomization Period through 24 Weeks (12 weeks in each Randomization Period)
Population: Participants who were randomized, received at least 1 dose of study drug after randomization, and had evaluable HE data during Randomization Periods.
Measure: Least Squares Mean (Standard Error); unit: events/participant/30 days
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 171 | 180
events/participant/30 days
  Total HE | 10.54 (0.67) | 10.37 (0.62)
  Nocturnal HE | 1.52 (0.13) | 1.34 (0.11)

3. Secondary Outcome: Percentage of Participants With Total and Nocturnal Hypoglycemic Events
Description: Total HE include any event based on a blood glucose <=70 mg/dL (3.9 mmol/L), with or without signs/symptoms of hypoglycemia or an event associated with signs/symptoms of hypoglycemia but without a glucose measurement. Nocturnal HE include any total HE that occurred between bedtime and waking. The percentage of participants was calculated by dividing the number of participants with hypoglycemic episodes by the total number of participants analyzed, multiplied by 100.
Time Frame: Baseline (Day 1) of Randomization Period through 24 weeks (12 weeks in each Randomization Period)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 171 | 180
percentage of participants
  Total HE | 98.2 | 97.8
  Nocturnal HE | 78.4 | 80.6

4. Secondary Outcome: Fasting Blood Glucose (FBG) Measured by Self-Monitored Blood Glucose
Description: FBG was measured by self-monitored blood glucose (SMBG). LS means were calculated using MMRM analysis including the following fixed effects: treatment, period, sequence, baseline FBG (last nonmissing value at or before randomization), baseline HbA1c (<=8.0% or >8.0%), week (defined from the start of each Randomization Period), and treatment-by-week interaction.
Time Frame: At 12 Weeks in Each Randomization Period
Population: Participants who were randomized, received at least 1 dose of study drug after randomization, and had evaluable FBG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 171 | 179
mg/dL | 131.35 (2.86) | 139.65 (2.87)

5. Secondary Outcome: Intra-Participant Variability of FBG at 12 Weeks
Description: FBG was measured by SMBG. Between-day glucose variability is measured by the standard deviation of FBG. LS means were calculated using MMRM analysis including the following fixed effects: treatment, period, sequence, baseline intra-participant variability in FBG (last nonmissing value at or before randomization), baseline HbA1c (<=8.0% or >8.0%), week (defined from the start of each Randomization Period), and treatment-by-week interaction.
Time Frame: At 12 Weeks in Each Randomization Period
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 171 | 179
mg/dL | 37.97 (1.73) | 39.80 (1.73)

6. Secondary Outcome: Fasting Serum Glucose (FSG) at 12 Weeks
Description: LS means for FSG (obtained from clinical laboratory tests) were calculated using MMRM analysis including the following fixed effects: treatment, period, sequence, baseline FSG (last nonmissing value at or before randomization), baseline HbA1c (<=8.0% or >8.0%), week (defined from the start of each Randomization Period), and treatment-by-week interaction.
Time Frame: At 12 Weeks in Each Randomization Period
Population: Participants who were randomized, received at least 1 dose of study drug after randomization, and had evaluable FSG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 171 | 177
mg/dL | 121.51 (4.27) | 120.45 (4.25)

7. Secondary Outcome: Change From Randomization to 12 Weeks in 9-Point SMBG
Description: SMBG measurements were taken at 9 time points: pre-morning meal, 2 hours post-morning meal, pre-midday meal, 2 hours post-midday meal, pre-evening meal, 2 hours post-evening meal, bedtime, at approximately 0300 hours, and the subsequent morning prior to the morning meal. SMBG measures were assessed at Weeks 0, 4, 8, and 12 within each Randomization Period. LS means were calculated using MMRM analysis including the following fixed effects: treatment, period, sequence, baseline SMBG (last nonmissing value at or before randomization), baseline HbA1c (<=8.0% or >8.0%), week (defined from the start of each Randomization Period), and treatment-by-week interaction.
Time Frame: Randomization, 12 Weeks in Each Randomization Period
Population: Participants who were randomized, received at least 1 dose of study drug after randomization, and had evaluable SMBG data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 164 | 169
mg/dL
  Pre-morning meal: number analyzed (Participants) | 163 | 168
  Pre-morning meal | -7.77 (3.79) | 0.07 (3.80)
  2 hours post-morning meal: number analyzed (Participants) | 163 | 167
  2 hours post-morning meal | -1.24 (4.03) | 8.13 (4.04)
  Pre-midday meal: number analyzed (Participants) | 164 | 168
  Pre-midday meal | 0.27 (3.55) | 14.87 (3.57)
  2 hours post-midday meal: number analyzed (Participants) | 164 | 167
  2 hours post-midday meal | 10.91 (3.93) | 5.40 (3.95)
  Pre-evening meal | 1.98 (3.81) | -1.34 (3.84)
  2 hours post-evening meal: number analyzed (Participants) | 163 | 167
  2 hours post-evening meal | 5.49 (4.06) | 8.33 (4.03)
  Bedtime: number analyzed (Participants) | 163 | 167
  Bedtime | 8.40 (4.15) | 5.36 (4.17)
  0300 hours: number analyzed (Participants) | 161 | 164
  0300 hours | -7.05 (3.55) | 4.71 (3.62)
  Subsequent morning pre-meal: number analyzed (Participants) | 162 | 167
  Subsequent morning pre-meal | -7.84 (3.20) | -2.44 (3.22)

8. Secondary Outcome: Self-Monitored Blood Glucose (SMBG) at 12 Weeks
Description: as for outcome 7
Time Frame: At 12 Week in Each Randomization Period
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 164 | 169
mg/dL
  Pre-morning meal: number analyzed (Participants) | 163 | 168
  Pre-morning meal | 133.21 (3.79) | 141.05 (3.80)
  2 hours post-morning meal: number analyzed (Participants) | 163 | 167
  2 hours post-morning meal | 151.03 (4.03) | 160.41 (4.04)
  Pre-midday meal: number analyzed (Participants) | 164 | 168
  Pre-midday meal | 122.96 (3.55) | 137.55 (3.57)
  2 hours post-midday meal: number analyzed (Participants) | 164 | 167
  2 hours post-midday meal | 147.05 (3.93) | 141.54 (3.95)
  Pre-evening meal | 137.75 (3.81) | 134.43 (3.84)
  2 hours post-evening meal: number analyzed (Participants) | 163 | 167
  2 hours post-evening meal | 150.37 (4.06) | 153.21 (4.03)
  Bedtime: number analyzed (Participants) | 163 | 167
  Bedtime | 153.81 (4.15) | 150.77 (4.17)
  0300 hours: number analyzed (Participants) | 161 | 164
  0300 hours | 131.40 (3.55) | 143.16 (3.62)
  Subsequent morning pre-meal: number analyzed (Participants) | 162 | 167
  Subsequent morning pre-meal | 125.16 (3.20) | 130.57 (3.22)

9. Secondary Outcome: Intra-participant Variability in SMBG at 12 Weeks
Description: A summary of glucose variability (intra-participant variability) as measured by the average of between-day standard deviations of individual SMBG time points. LS means were calculated using MMRM analysis including the following fixed effects: treatment, period, sequence, baseline intra-participant variability in SMBG (last nonmissing value at or before randomization), baseline HbA1c (<=8.0% or >8.0%), week (defined from the start of each Randomization Period), and treatment-by-week interaction.
Time Frame: At 12 Week in Each Randomization Period
Population: Participants who were randomized, received at least 1 dose of study drug after randomization, and had evaluable SMBG variability data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 154 | 153
mg/dL | 34.82 (1.30) | 36.21 (1.28)

10. Secondary Outcome: Change From Randomization to 12 Weeks in Body Weight
Description: LS means were calculated using MMRM analysis including the following fixed effects: treatment, period, sequence, baseline body weight (last nonmissing value at or before randomization), baseline HbA1c (<=8.0% or >8.0%), week (defined from the start of each Randomization Period), and treatment-by-week interaction.
Time Frame: Randomization, 12 Weeks in Each Randomization Period
Population: Participants who were randomized, received at least 1 dose of study drug after randomization, and had evaluable body weight data.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 170 | 177
kilograms (kg) | -0.06 (0.19) | 0.00 (0.19)

11. Secondary Outcome: Change From Day 1 of Lead-In Period to 36 Weeks in Body Weight
Description: LS means were calculated using MMRM analysis, including visit and baseline weight (last non-missing value at or before the beginning of Lead-in Period) as covariates.
Time Frame: Day 1 of Lead-In Period, 36 Weeks
Population: All enrolled participants who completed the first visit of the Lead-in Period, received at least 1 dose of study drug, and had evaluable body weight data.
Measure: Least Squares Mean (Standard Error); unit: kg
Groups:
- All Participants: All enrolled participants entered a 12-week lead-in period where they received fixed time dosing of LY2605541. Participants were then randomized to a fixed evening dose regimen or a variable time dose regimen for 12 weeks; after 12 weeks, they crossed over to the alternate regimen.
  Fixed-time dose regimen: Participant-specific dose of LY2605541 administered SQ at approximately the same time every evening for 12 weeks.
  Variable-time dose regimen: Participant-specific dose of LY2605541 administered SQ on a variable schedule (8- and 40-hour dosing intervals) for 12 weeks. Dosing schedules were to remain approximately the same throughout the 12 weeks.
Arm/Group | All Participants
Number analyzed (Participants) | 210
kg | -1.16 (0.29)

12. Secondary Outcome: Change From Randomization to 12 Weeks in HbA1c
Description: LS means were calculated using MMRM analysis including the following fixed effects: treatment, period, sequence, baseline HbA1c (last nonmissing value at or before randomization), week (defined from the start of each Randomization Period), and treatment-by-week interaction.
Time Frame: Randomization, 12 Weeks in Each Randomization Period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 171 | 180
percentage of HbA1c | 0.10 (0.04) | 0.18 (0.04)

13. Secondary Outcome: Participants With Treatment-Emergent Anti-LY2605541 Antibody Response
Description: The number of participants with a treatment emergent anti-LY2605541 antibody response (TEAR) is presented. Positive TEAR was defined as change from baseline to post-baseline in the anti-LY2605541 antibody level either from 1) undetectable to detectable or from 2) detectable to the value with at least 130% relative increase from baseline.
Time Frame: Day 1 of Lead-in Period through 36 Weeks
Population: Participants who completed the first visit of the Lead-in Period, received at least 1 dose of study drug, and had evaluable anti-LY2605541 antibody data.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 210
participants | 80

14. Secondary Outcome: Basal, Bolus, and Total Insulin Doses at 12 Weeks
Description: LS means were calculated using MMRM analysis including the following fixed effects: treatment, period, sequence, baseline insulin dose (last nonmissing value at or before randomization), baseline HbA1c (<=8.0% or >8.0%), week (defined from the start of each Randomization Period), and treatment-by-week interaction.
Time Frame: At 12 Weeks in Each Randomization Period
Population: Participants who were randomized, received at least 1 dose of study drug after randomization, and had evaluable insulin dose data.
Measure: Least Squares Mean (Standard Error); unit: units/kg/day
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 171 | 180
units/kg/day
  Basal | 0.50 (0.01) | 0.51 (0.01)
  Bolus | 0.20 (0.01) | 0.20 (0.01)
  Total Insulin | 0.71 (0.01) | 0.71 (0.01)

15. Secondary Outcome: Proportion of Bolus to Total Insulin Doses at 12 Weeks
Description: Proportion of bolus to total insulin dose is presented, where LS means were calculated using MMRM analysis including the following fixed effects: treatment, period, sequence, baseline proportion of bolus to total insulin dose (last nonmissing value at or before randomization), baseline HbA1c (<=8.0% or >8.0%), week (defined from the start of each Randomization Period), and treatment-by-week interaction.
Time Frame: At 12 Weeks in Each Randomization Period
Population: Participants who were randomized, received at least 1 dose of study drug after randomization, and had evaluable bolus to total insulin dose data.
Measure: Least Squares Mean (Standard Error); unit: units/day
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 171 | 178
units/day | 0.29 (0.01) | 0.28 (0.01)

16. Secondary Outcome: 0300-Hour Blood Glucose to Fasting Blood Glucose Excursion
Description: Excursion results were calculated by subtracting the 0300 hours glucose value from the next day pre-morning glucose value within a single SMBG profile. LS means were calculated using MMRM analysis including the following fixed effects: treatment, period, sequence, baseline 0300-hour to next day pre-breakfast excursion (last nonmissing value at or before randomization), baseline HbA1c (<=8.0% or >8.0%), week (defined from the start of each Randomization Period), and treatment-by-week interaction.
Time Frame: At 12 Week in Each Randomization Period
Population: Participants who were randomized, received at least 1 dose of study drug after randomization, and had evaluable SMBG excursion data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 158 | 162
mg/dL | -6.41 (3.64) | -15.24 (3.70)

17. Secondary Outcome: Change From Day 1 of Lead-in to 36 Weeks in Triglycerides, Total Cholesterol, Low-Density Lipoprotein Cholesterol (LDL-C), and High-Density Lipoprotein Cholesterol (HDL-C)
Description: LS means were calculated using MMRM analysis including visit and baseline lipid level (last nonmissing value at or before the beginning of Lead-in) as covariates.
Time Frame: Day 1 of Lead-In Period, 36 Weeks
Population: All enrolled participants who completed the first visit of the Lead-in Period, received at least 1 dose of study drug, and had evaluable lipid data.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 202
mg/dL
  Triglycerides: number analyzed (Participants) | 186
  Triglycerides | 26.44 (3.83)
  Total Cholesterol: number analyzed (Participants) | 186
  Total Cholesterol | 3.75 (1.91)
  LDL-C: number analyzed (Participants) | 181
  LDL-C | 4.45 (1.63)
  HDL-C: number analyzed (Participants) | 186
  HDL-C | -5.70 (0.82)

18. Secondary Outcome: Percentage of Participants With HbA1c <7.0% and ≤6.5% at 12 Weeks
Description: The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100.
Time Frame: At 12 Weeks in Each Randomization Period
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 Fixed Time Dosing | LY2605541 Variable Time Dosing
Number analyzed (Participants) | 167 | 167
percentage of participants
  HbA1c <7.0% | 60.5 | 54.5
  HbA1c <=6.5% | 34.1 | 34.1

ADVERSE EVENTS:
Groups:
- LY2605541 (All Participants): All participants who received at least 1 dose of LY2605541 during the Lead-In Period, Randomization Period 1, and Randomization Period 2.
Arm/Group | LY2605541 (All Participants) | LY2605541 Fixed Time Dosing, LY2605541 Variable Time Dosing | LY2605541 Variable Time Dosing, LY2605541 Fixed Time Dosing
Serious Adverse Events (participants affected / at risk) | 30/212 | 11/177 | 7/180
Other Adverse Events (participants affected / at risk) | 166/212 | 83/177 | 88/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 (All Participants) (N=212) | LY2605541 Fixed Time Dosing, LY2605541 Variable Time Dosing (N=177) | LY2605541 Variable Time Dosing, LY2605541 Fixed Time Dosing (N=180)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (3) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 24 (34) | 9 (9) | 6 (8)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemic seizure (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 (All Participants) (N=212) | LY2605541 Fixed Time Dosing, LY2605541 Variable Time Dosing (N=177) | LY2605541 Variable Time Dosing, LY2605541 Fixed Time Dosing (N=180)
Conjunctivitis (Eye disorders) | 2 (2) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 1 (1) | 1 (2)
Food poisoning (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (10) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 6 (7) | 1 (1) | 2 (2)
Fatigue (General disorders) | 4 (4) | 2 (2) | 3 (3)
Injection site pain (General disorders) | 3 (3) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 10 (23) | 1 (1) | 2 (2)
Local swelling (General disorders) | 3 (4) | 1 (1) | 3 (4)
Oedema peripheral (General disorders) | 3 (3) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 6 (6) | 2 (2) | 3 (3)
Gastroenteritis (Infections and infestations) | 9 (13) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 7 (7) | 4 (4) | 1 (1)
Hordeolum (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 13 (14) | 2 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 33 (47) | 11 (12) | 8 (8)
Sinusitis (Infections and infestations) | 11 (12) | 3 (3) | 5 (5)
Tooth infection (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 30 (33) | 9 (9) | 10 (10)
Urinary tract infection (Infections and infestations) | 5 (5) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 4 (5) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (2) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 2 (2) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 5 (5) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 5 (5) | 1 (1) | 2 (2)
Liver function test abnormal (Investigations) | 3 (3) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 6 (6) | 3 (3) | 3 (3)
Weight increased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3) | 2 (2)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 7 (10) | 2 (3) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 2 (2) | 2 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 2 (3) | 3 (3)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 5 (5) | 1 (1)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 10 (15) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days